CLINICAL TRIAL: NCT01045564
Title: Safety and Immunogenicity of GSK 15574484A Vaccine in Adults at Occupational Risk for Influenza A (H5N1) Exposure
Brief Title: Safety and Immunogenicity of Vaccine in Adults at Occupational Risk for Influenza A (H5N1) Exposure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was cancelled before enrolment for reasons not related to vaccine safety or efficacy.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: United States Department of Health and Human Services, Center for Disease Control and Prevention, National Institutes of Health, Department of Defense (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112576
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Influenza
Keywords: Immunogenicity; Vaccines; H5N1; Influenza; Pandemic; Human; Avian; Safety
MeSH Terms: conditions — Influenza, Human

ARMS (5):
- A (Experimental): One dose of study vaccine (GSK 1557484A) on Day 0, Day 182, and Day 364
  Interventions: Biological: GSK influenza virus H5N1 vaccine 1557484A
- B (Experimental): One dose of study vaccine (GSK 1557484A) on Day 0, Day 91, and Day 364
  Interventions: Biological: GSK influenza virus H5N1 vaccine 1557484A
- C (Experimental): One dose of study vaccine (GSK 1557484A) on Day 0, Day 21, and Day 364
  Interventions: Biological: GSK influenza virus H5N1 vaccine 1557484A
- D (Experimental): One dose of study vaccine (GSK 1557484A) on Day 0, Day 21, and Day 364
  Interventions: Biological: GSK influenza virus H5N1 vaccine 1557484A
- E (Experimental): One dose of study vaccine (GSK 1557484A) on Day 0, Day 21, and Day 364
  Interventions: Biological: GSK influenza virus H5N1 vaccine 1557484A

INTERVENTIONS:
Biological: GSK influenza virus H5N1 vaccine 1557484A — Three doses of GSK 1557484A administered intramuscularly (IM), the first and third in the deltoid region of the non-dominant arm and the second in the deltoid region of the dominant arm

SUMMARY:
The purpose of this study is to characterize the immunogenicity and safety of 3 doses of GSK's avian flu vaccine GSK 1557484A given at different time intervals to adults aged 18 years or greater who are at increased occupational risk of H5N1 exposure.

ELIGIBILITY:
Inclusion Criteria:

* A male or female 18 years of age or greater at the time of the first vaccination.
* At increased risk of occupational exposure to H5N1 influenza viruses based on:

  * Exposure to diseased poultry or wild birds,
  * Exposure, or potential exposure, to human cases of unidentified respiratory disease or known avian influenza,
  * Handling of human or avian microbiological specimens,
  * Handling of H5N1 viral isolates,
  * Or status critical to the implementation of emergency response measures in the event of an influenza pandemic declaration.
* Written informed consent obtained from the subject.
* Stable health status as defined by absence of a health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within one (1) month prior to enrollment.
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits.

Exclusion Criteria:

* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an oral temperature >= 37.8ºC, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Diagnosed with cancer, or treatment for cancer, within 3 years.

  * Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
  * Persons with a history of histologically-confirmed basal cell carcinoma of the skin successfully treated with local excision only are excepted and may enroll within 3 years of diagnosis, but other histologic types of skin cancer require a 3 year untreated and disease-free window as above.
  * Women who are disease-free 3 years or more after treatment for breast cancer and receiving long-term prophylactic tamoxifen are excepted and may enroll.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of systemic glucocorticoids within 1 month prior to study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrollment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination, are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine.
* Administration of any vaccines within 30 days before any study vaccination.
* Exposure to any investigational or non-registered product (drug or vaccine) during this trial, or within 30 days prior to study enrollment. Potential subjects in the follow-up (i.e., no treatment) phase of a prior investigational study may be enrolled if the investigator's judgment is that it will have no effect on safety, reactogenicity, or immunogenicity endpoints in this study; and that it does not violate the protocol requirements of the prior trial.
* Any known or suspected allergy to any constituent of influenza vaccines (including egg proteins or mercurial preservatives); a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Receipt of analgesic or antipyretic medication with the specific intent of prophylaxis of vaccine reactogenicity on the day of treatment constitutes a contraindication to administration of study vaccine at that point in time;
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result prior to any vaccination.
* Lactating or nursing.
* Women of child bearing potential who lack a history of reliable contraceptive practices. The provision of this history does NOT replace the requirement to perform, and obtain negative results in pregnancy urine tests prior to treatments.

  * Reliable contraceptive practices include:
  * consistent abstinence from heterosexual activity,
  * consistent use of combined or progestogen oral contraceptives,
  * injectable progestogen,
  * implants of levonorgestrel,
  * estrogen or estrogen/ progestogen vaginal ring,
  * percutaneous contraceptive patches or intrauterine device (IUD) or intrauterine system (IUS),
  * vasectomy with documented azoospermia of >= 6 months of the sole male partner, or
  * double barrier method (condom or occlusive cap plus spermicidal agent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Booster humoral immune response in terms of Hemagglutination Inhibition (HI) antibodies (after second vaccination). | Day 0 and 21 days after the second vaccination

SECONDARY OUTCOMES:
Booster humoral immune response in terms of Hemagglutination Inhibition (HI) antibodies.on secondary readouts (after second vaccination) | Days 0 and 21 days after second vaccination
Primary humoral immune response in terms of Hemagglutination Inhibition (HI) antibodies (after first vaccination) | Days 0, 21 and 42 after first vaccination (depending on vaccination schedule)
Humoral immune response in terms of Hemagglutination Inhibition (HI) antibodies (after third vaccination) | Days 364, 385, and 546
Humoral immune response in terms of microneutralization titers and cellular T-cell immune response | Days 0, 21, 21 days after second vaccination, 364, 385, and 546 (depending on vaccination schedule)
Occurrence of specifically-solicited local and general signs and symptoms | During a 7-day follow up period after each vaccine dose
Occurrence of all unsolicited adverse events | During a 21-day follow up period after each vaccine dose
Occurrence of serious adverse events and adverse events of special interest | From day 0 through day 546

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Silver Spring, Maryland